CLINICAL TRIAL: NCT04647344
Title: An Open-label, Multicenter, Phase Ib/II Study of AK104, Combined Chemotherapy as First-line Therapy to Treat Locally Advanced or Metastatic Non-small Cell Lung Carcinoma
Brief Title: A Study of AK104 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-207
Record Dates: First submitted 2020-11-21; First posted 2020-11-30 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer Non-Small Cell Stage IIIB/IIIC/IV
MeSH Terms: interventions — Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nonsquamous NSCLC (Experimental)
  Interventions: Drug: AK104 plus Carboplatin and Pemetrexed
- Squamous NSCLC (Experimental)
  Interventions: Drug: AK104 plus Carboplatin and paclitaxel

INTERVENTIONS:
Drug: AK104 plus Carboplatin and Pemetrexed — Subjects receive AK104 15mg/kg intravenously (IV) plus pemetrexed 500 mg/m^2 IV and carboplatin area under the curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK104 15mg/kg IV plus pemetrexed 500 mg/m^2 IV Q3W until progression.
  Arms: Nonsquamous NSCLC
Drug: AK104 plus Carboplatin and paclitaxel — Subjects receive AK104 15mg/kg intravenously (IV) plus paclitaxel 175 mg/m^2 IV and carboplatin area under the curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by AK104 15mg/kg IV IV Q3W until progression.
  Arms: Squamous NSCLC

SUMMARY:
This is a phase Ib/II , open-label, multicenter single arm study designed to evaluate the efficacy, safety, tolerability, pharmacokinetic (PK), and immunogenicity of AK104 combined with Carboplatin and Pemetrexed/ Paclitaxel as first-line therapy in patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the informed consent form.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Expected life expectance ≥ 3 months.
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC.
* No prior systemic chemotherapy for advanced or metastatic NSCLC. Subjects who have received prior adjuvant chemotherapy or neoadjuvant chemotherapy with curative intent, or definitive chemoradiotherapy for advanced disease, will be eligible provided that progression has occurred >6 months from last treatment.
* At least one measurable tumor lesion per RECIST 1.1 criteria. A lesion previously irradiated will not be considered a target lesion.
* Subjects must provide an available tumor tissue sample taken < 1 year prior to first dose of study treatment.
* Subjects must provide wild-type epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) reported by tissue-based tests（for non-squamous NSCLC subjects only）.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.

Key Exclusion Criteria:

* Subjects who are diagnosed as NSCLC that harbors an epidermal growth factor receptor (EGFR)-sensitizing mutation or anaplastic lymphoma kinase (ALK) gene translocation.
* Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the subject is ineligible
* Received prior treatment with EGFR inhibitors or ALK inhibitors.
* Is currently participating intervention study or has participated in a study of an investigational agent or investigational device within 4 weeks prior to administration of AK104.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as Inducible T-cell co-stimulator (ICOS) or agonists (e.g. CD40, CD137, GITR and OX40 etc).
* Subjects who received non-thoracic radiotherapy >30 Gy within 4 weeks prior to the first dose , or thoracic radiotherapy >30 Gy within 24 weeks prior to the first dose study drug.
* Other active malignancies within 2 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease,
* Subjects who require systemic corticosteroids (a dose equivalent to >10 mg/day prednisone) or other immunosuppressive drugs within 14 days prior to administration of AK104.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
* Known history of active tuberculosis (TB).
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 1000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <1000 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Presence of meningeal metastasis, spinal cord compression, leptomeningeal disease or active brain metastasis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria, with the exception of alopecia.
* Receipt of live vaccination within 30 days of planned treatment start, or plan to receive live vaccine during the study.
* Known history of server hypersensitivity to other monoclonal antibodies.
* Known severe allergic reactions to pemetrexed, paclitaxel, carboplatin or platinum-containing component, or their preventive medications.
* Known allergic reactions to any ingredients of AK104.
* Known history of substance abuse, or alcohol abuse
* Pregnant or lactating women.
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing adverse events (AEs) (Phase Ib) | From the time of informed consent through 90 days following termination of treatment with investigational product
Objective response rate (ORR) assessed by investigator | Up to 2 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
Duration of response (DoR) | Up to 2 years
Progression-free survival (PFS) | Up to 2 years
Overall survival (OS) | Up to 2 years
Time to response (TTR) | Up to 2 years
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of AK104 through 90 days after last dose of AK104
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University Cancer Center, Guangzhou, China
Locations (1):
- Sun Yat-Sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No